CLINICAL TRIAL: NCT06084247
Title: An Open Label Randomized-control Study on the Efficacy of the KARL STORZ Curved Fetoscope (11508aak) and Its Straight Version (11506aak) for Laser Photocoagulation of Placental Anastomoses
Brief Title: The Efficacy of the KARL STORZ Curved Fetoscope and Straight Fetoscope for Laser Photocoagulation of Placental Anastomoses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jimmy Espinoza (Other)
Responsible Party: Sponsor-Investigator, Jimmy Espinoza, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0622
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Twin to Twin Transfusion Syndrome
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- KARL STORZ Curved Scope (Experimental)
  Interventions: Device: Curved KARL STORZ fetoscope
- Conventional scopes (Active Comparator)
  Interventions: Device: Conventional Scopes

INTERVENTIONS:
Device: Curved KARL STORZ fetoscope — The KARLZ STORZ curved scope is used to see the inside of a pregnant person's uterus during minimally invasive surgery, similar to conventional scopes. The curved scope is rounded and thought to help visualize the anterior placenta because of its position on the uterus.
  Arms: KARL STORZ Curved Scope
Device: Conventional Scopes — The conventional scopes are regularly used during laser photocoagulation of placental anastomoses.
  Arms: Conventional scopes

SUMMARY:
The purpose of this study is to evaluate the efficacy of KARL STORZ curved fetoscope (11508AAK) and its straight version (11506AAK) for laser photocoagulation of placental anastomoses in patients with an anterior placenta and Twin to Twin Transfusion Syndrome (TTTS).

ELIGIBILITY:
Inclusion Criteria:

* pregnancy
* The patient fulfills the criteria for laser photocoagulation of placental anastomoses based on the standard of care
* fetal diagnosis of twin-to-twin transfusion syndrome
* Anterior placenta
* The patient provides signed informed consent that details the maternal and fetal risks involved with the procedure

Exclusion Criteria:

* Contraindication to abdominal surgery, fetoscopic surgery, or general anesthesia
* Allergy or previous adverse reaction to a study medication specified in this protocol
* The patient does not fulfill the conventional criteria to undergo in-utero surgery, which is specific for each surgery
* Preterm labor, preeclampsia, or a uterine anomaly (e.g., large fibroid tumor) that is unavoidable during surgery in the index pregnancy
* Fetal aneuploidy, genomic variants of known significance if an amniocentesis has been performed, other major fetal anomalies or disorders that may impact the fetal/neonatal survival, or a known syndromic mutation
* Suspicion of a major recognized syndrome by ultrasound or MRI
* Maternal BMI >40 kg/m2
* High risk for fetal hemophilia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Operative time in minutes | during surgery
  Time from from operative cannula insertion until it is removed

SECONDARY OUTCOMES:
Number of Participants that have a gestational age of less than 37 weeks | at time of delivery (about 20 weeks from surgery)
Number of times additional fetoscopes are entered into the amniotic cavity to confirm completion of the in-utero intervention | end of surgery (about 60 minutes after start of surgery)
Total number of procedures with completion of the laser ablation | end of surgery (about 60 minutes after start of surgery)
Improved visualization as assessed by the Likert scale | end of surgery (about 60 minutes after start of surgery)
  This is reported categorically as strongly disagree, disagree, neither agree not disagree, agree and strongly agree. This is not a validated scale and does not have an official title. The minimum value is strongly disagree and the maximum value is strongly agree. Higher scores mean better outcomes.
Improved angle for laser visualization as assessed by the Likert scale | end of surgery (about 60 minutes after start of surgery)
  This is reported categorically as strongly disagree, disagree, neither agree not disagree, agree and strongly agree
Total number of fetuses alive, after the laser photocoagulation procedure | at discharge from hospital (about 24 hours after surgery)
Total number of maternal patients that present with morbidity | at discharge from hospital (about 24 hours after surgery)
Total number of patients that have maternal and/or fetal perioperative complications | end of surgery (about 60 minutes after start of surgery)
The number of participants that develop twin-anemia-polycythemia sequence (TAPS) | end of surgery (about 60 minutes after start of surgery)
Number of live births | at time of delivery (about 20 weeks from surgery)
Number of neonates with a short-term morbidity | from birth until hospital discharge
Infant development score using the Ages & Stages Questionnaires, Third Edition (ASQ-3) | 24 months of age
  Scored items on ASQ-3 address 5 areas of child development: communication, gross motor, Fine motor, problem solving, and personal-social and each of these have 6 questions each and is scored as yes( 10 points), sometimes (5 points) and not yet (0 points)-the total score is calculated for each area and scores should fall between 0-60, and a higher score indicates more development.
  There is a 9 item overall developmental section that is answered categorically as yes or no answer

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Espinoza, MD, MSc,FACOG, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No